CLINICAL TRIAL: NCT00934427
Title: A Study of a Topical Formulation of Nitroglycerin, Vascana® (MQX-503), and Matching Vehicle in the Treatment and Prevention of Symptoms Associated With Raynaud's Phenomenon
Brief Title: Study of a Topical Formulation for the Treatment and Prevention of Raynaud's Phenomenon Symptoms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MediQuest Therapeutics (Industry)
Responsible Party: Jeff Gregory, MD / Medical Director, MediQuest Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-001
Record Dates: First submitted 2009-06-26; First posted 2009-07-08 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Raynaud Disease
Keywords: Raynaud's; scleroderma; nitroglycerin; MQX-503; treatment
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vascana (Active Comparator)
  Interventions: Drug: 0.9% nitroglycerin in TAM cream
- Vehicle (Placebo Comparator)
  Interventions: Drug: vehicle cream

INTERVENTIONS:
Drug: 0.9% nitroglycerin in TAM cream — 0.5 g of Vascana (0.9% nitroglycerin in proprietary vehicle cream) is applied topically BID for one day before certain planned cold exposures, once just before same planned cold exposures, and, if needed, right after the start of symptoms during same planned cold exposures
  Other Names: Vascana
  Arms: Vascana
Drug: vehicle cream — 0.5g of vehicle cream is topically administered BID for one day before certain planned cold exposures, once just before certain planned cold exposures, and, if needed, right after the start of symptoms during certain planned cold exposures
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine if Vascana, a novel topical formulation of nitroglycerin, is effective in the treatment and prevention of the symptoms associated with Raynaud's Phenomenon.

DETAILED DESCRIPTION:
Raynaud's Phenomenon is a sometimes debilitating condition in which blood flow to the fingers or toes is compromised when a patient is exposed to cold or stress. Current therapies for Raynaud's are suboptimal because they are associated with significant side effects. In this study, patient responses to cold temperature exposures in a climate-controlled room after application of the study medication are measured.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Raynaud's phenomenon as determined by a history of cold sensitivity with pain, numbness, and/or tingling along with pallor or cyanosis of the fingers
* a history of at least two Raynaud's events during a typical winter day
* must be willing to apply creams to fingers
* must be willing to undergo cold temperature exposure
* must be willing and able to stop certain medications
* must be willing to use effective contraception, if applicable

Exclusion Criteria:

* had a Raynaud's attack that required hospital or clinic intervention
* has allergies to nitroglycerin or topical medication ingredients
* has a history of migraine or chronic pain
* has an unstable medical problem that could interfere with the study
* had a heart attack or uncontrolled heart problems, hypertension, or hypotension in the past 3 months
* used any investigational drug in the past 4 weeks
* has significantly abnormal laboratory tests
* had certain major surgeries in the past 6 months
* has skin lesions on certain parts of the fingers
* women who are pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Response rate as measured by changes in severity of the Raynaud's symptom most bothersome to the individual patient (Pain, Numbness, or Tingling) | 2 weeks

SECONDARY OUTCOMES:
Changes from baseline in severity of each Raynaud's symptom (Pain, Numbness, and Tingling) | 2 weeks
Changes from baseline in duration of Raynaud's attacks | 2 weeks
Changes from baseline in number of Raynaud's attacks | 2 weeks
Changes from baseline in the Raynaud's Condition Score | 2 weeks
Changes in the maximum reduction in skin temperature | 2 weeks
Changes from baseline in overall disease severity measures | 2 weeks
Changes in the time to return to baseline skin temperature | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Gregory, MD, Study Director — MediQuest Therapeutics
Locations (11):
- United States (11):
  - Stanford University, Redwood City, California
  - University of Connecticut, Farmington, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Medicine and Dentistry in New Jersey, New Brunswick, New Jersey
  - Carolina Arthritis, Wilmington, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin